CLINICAL TRIAL: NCT03159702
Title: Propylene Glycol-Free Melphalan HCl (EVOMELA®) in Combination With Fludarabine and Total Body Irradiation Based Reduced Intensity Conditioning for Haploidentical Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Mehdi Hamadani, Professor, Department of Medicine, Division of Hematology/Oncology, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO29507
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Results first posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Hematological Malignancy; Multiple Myeloma
Keywords: hematological malignancy; EVOMELA; Melphalan HCl; Total Body Irradiation; Reduced Intensity Conditioning; Haploidentical Transplantation; Fludarabine; Hematologic Diseases
MeSH Terms: conditions — Hematologic Neoplasms; Multiple Myeloma; Hematologic Diseases | interventions — Melphalan; fludarabine; fludarabine phosphate; Whole-Body Irradiation

STUDY DESIGN:
Intervention Model Description: Study subjects will receive different doses of Melphalan during the trial. This is done for safety per FDA recommendations. Subjects younger than 60 years or have will receive doses at 140 mg/m^2/day while subject 60 years or old or have a Hematopoietic Cell Transplant-Co-morbidity Index (HCT-CI) score of >3 will receive 70 mg/m^2/day. The populations will be combined for analysis and reporting.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- MEL/FLU and Total-Body Irradiation (TBI) (Experimental): For patients who are < 60 years.
  * Melphalan: 140 mg/m2/day IV on Day: -6
  * Fludarabine: 40 mg/ m2/day IV Days: -5 -4, -3, -2 (Adults: creatinine clearance (CrCl) may be estimated by the Cockcroft Formula: CrCl = [(140-age) x weight (kg) x 0.85 (for women only)]/ [72 x creat (mg/dl)].)
  * TBI: 200 cGy Day: -1.
  For patients who are ≥60 years and/or Hematopoietic Cell Transplant-Co-morbidity Index (HCT-CI) score of >3 (at the discretion of treating physician will have an option to receive):
  * Melphalan: 70 mg/m2/day IV on Day -6.
  * Fludarabine: 40 mg/m2/day IV Days -5, -4, -3, -2.
  * TBI: 200 cGy; Days -1.
  Interventions: Drug: Evomela; Drug: Fludarabine; Radiation: Total Body Irradiation; Other: Haploidentical Hematopoietic Cell Transplantation

INTERVENTIONS:
Drug: Evomela — 140 mg/m^2/day IV on Day -6 for patients who are < 60 years of age. 70 mg/m^2/day IV on Day -6 For patients who are ≥60 years or have a HCT-CI score of >3
  Other Names: Melphalan
Drug: Fludarabine — 40 mg/ m^2/day intravenous on Days: -5 -4, -3, -2
  Other Names: Fludara
Radiation: Total Body Irradiation — 200 cGy on Day: -1
Other: Haploidentical Hematopoietic Cell Transplantation — This is a procedure that uses healthy blood-forming cells from a half-matched donor, typically a family member, to replace a patient's unhealthy ones.

SUMMARY:
This is an open-label, single-arm, phase II study to determine the safety of propylene glycol-free melphalan HCl (EVOMELA®), in combination with fludarabine and total-body irradiation-based reduced-intensity conditioning for haploidentical transplantation. In addition, the study evaluates the one-year progression-free survival of patients undergoing this treatment.

DETAILED DESCRIPTION:
OVERVIEW:

Elderly and infirm patients with hematological malignancies often cannot undergo allogeneic hematopoietic cell transplantation (HCT) because of high-toxicity rates and nonrelapse mortality (NRM) associated with higher-intensity conditioning allografts.

Reduced-intensity conditioning (RIC) transplantation has emerged as an attractive alternative for these populations.

FLUDARABINE/MELPHALAN. In RIC, fludarabine is often used as the lymphocyte-depleting component to facilitate donor-cell engraftment. This drug can be given once daily because of its plasma half-life. M.D. Anderson pioneered the use of fludarabine melphalan (FLU/MEL) conditioning, which has since gained wide usage. (1) Melphalan is convenient, has broad antitumor activity in hematologic malignancies and has immunosuppressive effects. The Flu/Mel conditioning regimen can provide long-term disease control, especially in the subset of patients with chemo sensitive disease. (1) TOTAL-BODY IRRADIATION. In a recent study, total-body irradiation (200 cGy) was used with flu/mel for advanced lymphoma treated with HCT. With a median follow-up time close to two years, the survival of these mostly advanced, relapsed/refractory patients was very encouraging with overall survival of 54% and progression-free survival of 54% for the entire group. (2) Treatment-related mortality was low at day 100 (9.1%) and two years (19%) after transplantation, with stable engraftment achieved in the great majority of patients.

PROPYLENE GLYCOL-FREE MELPHALAN HCL (EVOMELA®). In theory, intensifying the dose of melphalan in flu/mel conditioning could provide better disease control post HCT, allowing more time for curative graft-versus-leukemia effects to emerge. The use of the commercial formulation of melphalan (Alkeran®) proved somewhat problematic, however, because it must be reconstituted with propylene glycol, a substance that has been associated with toxic side effects. The substitution of Captisol® in propylene glycol-free melphalan HCl (EVOMELA®) for Injection (Spectrum Pharmaceuticals, Inc.) for the excipients found in Alkeran®, directly overcomes the formulation limitations noted with Alkeran®.

STUDY RATIONALE. The preliminary data suggest that the substitution of Captisol® in EVOMELA® for the excipients found in Alkeran® directly overcomes the formulation limitations and provides a potentially safer melphalan formulation for administration at higher doses used in HCT conditioning regimens.

Based on these observations, we now propose a phase II study of a RIC regimen consisting of EVOMELA® in combination with fludarabine and total-body irradiation for patients undergoing haplo-HCT. The study will investigate the safety and tolerability of this conditioning approach. While the FDA indication for EVOMELA® is for myeloablative conditioning prior to autologous HCT in patients with multiple myeloma, we anticipate our study will provide critical preliminary data to explore this formulation in allogeneic HCT conditioning.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of hematological malignancy undergoing a related donor haploidentical HCT.*
* Patients aged ≥18 are eligible.
* Bilirubin ≤ 2 x the upper limit of normal (ULN). For patients with Gilbert's syndrome or suspected mild veno-occlusive disease, bilirubin ≤ 3 x ULN is permitted.
* Adequate renal function as defined by a serum creatinine clearance of > 30 mL/min calculated by Cockcroft-Gault equation.
* Left ventricular ejection fraction ≥40%. No uncontrolled arrhythmias or New York Heart Association class III-IV heart failure.
* Forced expiratory volume (FEV1) or diffusion capacity for carbon monoxide (DLCO) corrected for hemoglobin ≥ 50% of predicted.
* Karnofsky performance status > 60.
* Graft source of peripheral blood (the infused cluster of differentiation 34 (CD34)+ cell dose will be capped at 5 x 10^6 CD34+ cells/kg recipients actual body weight) or bone marrow (the ideal infused total nucleated cell dose (TNC) will be targeted at 4 x 10^8/kg recipient actual body weight).
* A negative pregnancy test will be required for all women of child bearing potential. Females of child bearing potential should agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug and must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, or agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.). Breast-feeding is not permitted.
* Male patients, even if surgically sterilized (i.e., status post-vasectomy), must agree to one of the following: practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, or must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, or agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
* No evidence of uncontrolled bacterial, viral or fungal infections at the time of enrollment.
* Transplant recipient able to give informed consent. * Patients must be human leukocyte antigen (HLA) typed at high resolution using DNA based typing at the following HLA loci: HLA-A, -B, -C and DRB1 and have available: A related haploidentical bone marrow donor with two, three or four HLA-mismatches. A unidirectional mismatch in either the graft-versus-host or host-versus-graft direction is considered a mismatch. The donor and recipient must be HLA identical for at least one antigen (using high-resolution DNA-based typing) at the following genetic loci: HLA-A, HLA-B, HLA-C, and HLA-DRB1. Fulfillment of this criterion shall be considered sufficient evidence that the donor and recipient share one HLA haplotype, and typing of additional family members is not required.

Exclusion Criteria:

* Patient must not have a healthy, eligible and readily available HLA-identical sibling donor or a volunteer adult unrelated donor (matched at allele-level at HLA-A, -B, -C and -DRB1).
* No serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.\
* Presence of active disease in acute myeloid leukemia (AML)/myelodysplastic syndrome (MDS): patients with active disease defined as >5% blasts in bone marrow and/or circulating leukemic blasts in peripheral blood, patients with known active central nervous disease involvement with leukemia/lymphoma or lymphoma patients with progressive disease on clinical and/or radiographic assessment are not eligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2025-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Hamadani, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Besien K, Devine S, Wickrema A, Jessop E, Amin K, Yassine M, Maynard V, Stock W, Peace D, Ravandi F, Chen YH, Hoffman R, Sossman J. Regimen-related toxicity after fludarabine-melphalan conditioning: a prospective study of 31 patients with hematologic malignancies. Bone Marrow Transplant. 2003 Sep;32(5):471-6. doi: 10.1038/sj.bmt.1704166. PMID 12942092
- [Background] Brammer JE, Khouri I, Gaballa S, Anderlini P, Tomuleasa C, Ahmed S, Ledesma C, Hosing C, Champlin RE, Ciurea SO. Outcomes of Haploidentical Stem Cell Transplantation for Lymphoma with Melphalan-Based Conditioning. Biol Blood Marrow Transplant. 2016 Mar;22(3):493-8. doi: 10.1016/j.bbmt.2015.10.015. Epub 2015 Oct 20. PMID 26497906

RESULTS

PARTICIPANT FLOW:
Groups:
- MEL/FLU and Total-Body Irradiation (TBI): For patients who are < 60 years.
  * Melphalan: 140 mg/m2/day IV on Day: -6
  * Fludarabine: 40 mg/ m2/day IV Days: -5 -4, -3, -2 (Adults: creatinine clearance (CrCl) may be estimated by the Cockcroft Formula: CrCl = [(140-age) x weight (kg) x 0.85 (for women only)]/ [72 x creat (mg/dl)].)
  * TBI: 200 cGy Day: -1.
  For patients who are ≥60 years and/or Hematopoietic Cell Transplant-Co-morbidity Index (HCT-CI) score of >3 (at the discretion of treating physician will have an option to receive):
  * Melphalan: 70 mg/m2/day IV on Day -6.
  * Fludarabine: 40 mg/m2/day IV Days -5, -4, -3, -2.
  * TBI: 200 cGy; Days -1.
  Evomela: 140 mg/m^2/day IV on Day -6 for patients who are < 60 years of age. 70 mg/m^2/day IV on Day -6 For patients who are ≥60 years or have a HCT-CI score of >3
  Fludarabine: 40 mg/ m^2/day intravenous on Days: -5 -4, -3, -2
  Total Body Irradiation: 200 cGy on Day: -1
Period: Overall Study
Arm/Group | MEL/FLU and Total-Body Irradiation (TBI)
Started | 43
Completed | 43
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MEL/FLU and Total-Body Irradiation (TBI)
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 36
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) of Participants With Hematological Malignancies Undergoing Treatment.
Description: Progression-free survival (PFS) is defined as the interval from the date of transplantation to the earlier of the following events: (1) the first documented objective disease progression; (2) death from any cause. Subjects without documented PD/death will be censored at the earliest of the of the following times: (1) the starting time of a new treatment other than the study treatment; (2) the last efficacy assessment date.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Groups:
- MEL/FLU and Total-Body Irradiation (TBI): For patients who are < 60 years.
  * Melphalan: 140 mg/m2/day IV on Day: -6
  * Fludarabine: 40 mg/ m2/day IV Days: -5 -4, -3, -2 (Adults: creatinine clearance (CrCl) may be estimated by the Cockcroft Formula: CrCl = [(140-age) x weight (kg) x 0.85 (for women only)]/ [72 x creat (mg/dl)].)
  * TBI: 200 cGy Day: -1.
  For patients who are ≥60 years and/or Hematopoietic Cell Transplant-Co-morbidity Index (HCT-CI) score of >3 (at the discretion of treating physician will have an option to receive):
  * Melphalan: 70 mg/m2/day IV on Day -6.
  * Fludarabine: 40 mg/m2/day IV Days -5, -4, -3, -2.
  * TBI: 200 cGy; Days -1.
  Evomela: 140 mg/m^2/day IV on Day -6 for patients who are < 60 years of age. 70 mg/m^2/day IV on Day -6 For patients who are ≥60 years or have a HCT-CI score of >3
  Fludarabine: 40 mg/ m^2/day intravenous on Days: -5 -4, -3, -2
  Total Body Irradiation: 200 cGy on Day: -1
  Haploidentical Hematopoietic Cell Transplantation: This is a procedure that uses healthy blood-forming cells from a half-matched donor, typically a family member, to replace a patient's unhealthy ones.
Arm/Group | MEL/FLU and Total-Body Irradiation (TBI)
Number analyzed (Participants) | 43
Participants | 17

2. Primary Outcome: Serious Adverse Events (SAE).
Description: An SAE is defined as any untoward medical occurrence at any dose, including death, life threatening, hospitalization, disability/incapacity, medically important event. The measure of this outcome is the number of participants with SAEs.
Time Frame: 2 Years
Measure: Count of Participants; unit: Participants
Arm/Group | MEL/FLU and Total-Body Irradiation (TBI)
Number analyzed (Participants) | 43
Participants | 12

3. Secondary Outcome: Nonrelapse Mortality Rate.
Description: This is the number of participants expiring without recurrent or progressive disease after transplantation.
Time Frame: 1 Year
Reporting Status: Not Posted, anticipated posting 2026-12

4. Secondary Outcome: Overall Survival
Description: The number of participants still alive at one year and 2 years.
Time Frame: 1 Year and 2 Year
Reporting Status: Not Posted

5. Secondary Outcome: Number of Subjects With Relapse of Disease.
Description: The number of participants who relapse following reduced-intensity conditioning haploidentical transplantation at Day 100 and 1 Year.
Time Frame: Day 100 and 1 Year
Reporting Status: Not Posted

6. Secondary Outcome: Neutrophil Recovery
Description: The average of the number of days that it takes for neutrophil recovery from reduced-intensity conditioning haploidentical transplantation. Neutrophil recovery means absolute neutrophil count of 0.5x10^3 cells/uL.
Time Frame: Day 30
Reporting Status: Not Posted

7. Secondary Outcome: Platelet Recovery
Description: The average of the number of days that it takes for platelet recovery from reduced-intensity conditioning haploidentical transplantation. Platelet recovery means absolute neutrophil count of 50x10^3 cells/uL.
Time Frame: Day 30
Reporting Status: Not Posted

8. Secondary Outcome: Acute Graft-versus-host Disease (GVHD) at Day 100 and 180.
Description: The number of participants with graft-versus-host disease using the Center for International Bone Marrow Transplant Research criteria.
Time Frame: Days 100 and 180
Reporting Status: Not Posted

9. Secondary Outcome: Rates of Chronic GVHD at One-year Post Transplantation.
Description: The number of participants with chronic GVHD at one-year post transplantation using the Center for International Bone Marrow Transplant Research criteria.
Time Frame: 1 Year
Reporting Status: Not Posted

10. Secondary Outcome: Primary Graft Failure
Description: Number of subjects whose grafts failed to implant.
Time Frame: Day 30
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 Years
Arm/Group | MEL/FLU and Total-Body Irradiation (TBI)
All-Cause Mortality (participants affected / at risk) | 18/43
Serious Adverse Events (participants affected / at risk) | 12/43
Other Adverse Events (participants affected / at risk) | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEL/FLU and Total-Body Irradiation (TBI) (N=43)
CMV Viremia (Infections and infestations) | 1 (1)
HHVS Virus (Infections and infestations) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Cytokine release syndrome (Immune system disorders) | 2 (2)
Upper respiratory infection (Infections and infestations) | 1 (1)
Cervical Mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Sepsis (Infections and infestations) | 3 (3)
Neoplasms benign, malignant and unspecified (incl cysts and polys) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Typhlitis (Gastrointestinal disorders) | 1 (1)
Altered mental status (Nervous system disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Blood in stool (Gastrointestinal disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEL/FLU and Total-Body Irradiation (TBI) (N=43)
Abdominal pain (Gastrointestinal disorders) | 17 (33)
Acute kidney injury (Renal and urinary disorders) | 7 (16)
Alanine aminotransferase increased (Investigations) | 8 (16)
Alkaline phosphatase increased (Investigations) | 4 (13)
Anal pain (Gastrointestinal disorders) | 5 (6)
Anemia (Blood and lymphatic system disorders) | 31 (87)
Anorexia (Metabolism and nutrition disorders) | 20 (42)
Aspartate aminotransferase increased (Investigations) | 8 (18)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9)
Bladder spasm (Renal and urinary disorders) | 6 (6)
Chills (General disorders) | 12 (18)
Constipation (Gastrointestinal disorders) | 15 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (10)
Creatinine increased (Investigations) | 18 (37)
Diarrhea (Gastrointestinal disorders) | 38 (86)
Dysgeusia (Nervous system disorders) | 5 (8)
Dyspepsia (Gastrointestinal disorders) | 8 (8)
Dysphagia (Gastrointestinal disorders) | 7 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 18 (31)
Edema limbs (General disorders) | 20 (28)
Electrocardiogram QT corrected interval prolonged (Investigations) | 5 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 (12)
Fatigue (General disorders) | 28 (55)
Febrile neutropenia (Blood and lymphatic system disorders) | 25 (32)
Fecal incontinence (Gastrointestinal disorders) | 13 (20)
Fever (General disorders) | 22 (37)
Flushing (Vascular disorders) | 6 (7)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 6 (9)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 8 (9)
Hallucinations (Psychiatric disorders) | 4 (4)
Headache (Nervous system disorders) | 20 (38)
Hematuria (Renal and urinary disorders) | 12 (15)
Hemorrhoids (Gastrointestinal disorders) | 11 (11)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 13 (23)
Hyperkalemia (Metabolism and nutrition disorders) | 10 (21)
Hypertension (Vascular disorders) | 21 (61)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 6 (12)
Hypoalbuminemia (Metabolism and nutrition disorders) | 24 (47)
Hypocalcemia (Metabolism and nutrition disorders) | 26 (70)
Hypokalemia (Metabolism and nutrition disorders) | 27 (71)
Hypomagnesemia (Metabolism and nutrition disorders) | 30 (49)
Hyponatremia (Metabolism and nutrition disorders) | 23 (54)
Hypophosphatemia (Metabolism and nutrition disorders) | 23 (46)
Hypotension (Vascular disorders) | 19 (54)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8 (14)
Insomnia (Psychiatric disorders) | 12 (20)
Lymphocyte count decreased (Investigations) | 30 (66)
Mucositis oral (Gastrointestinal disorders) | 17 (23)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Nausea (Gastrointestinal disorders) | 37 (72)
Neutrophil count decreased (Investigations) | 31 (107)
Non-cardiac chest pain (General disorders) | 5 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (10)
Pericardial effusion (Cardiac disorders) | 4 (5)
Platelet count decreased (Investigations) | 35 (167)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Proteinuria (Renal and urinary disorders) | 4 (13)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13 (18)
Dysuria (Renal and urinary disorders) | 4 (5)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Sinus tachycardia (Cardiac disorders) | 17 (35)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 9 (16)
Tremor (Nervous system disorders) | 6 (9)
Urinary frequency (Renal and urinary disorders) | 12 (18)
Urinary incontinence (Renal and urinary disorders) | 11 (13)
Urinary urgency (Renal and urinary disorders) | 6 (8)
Vomiting (Gastrointestinal disorders) | 19 (36)
Weight gain (Investigations) | 4 (11)
Weight loss (Investigations) | 7 (7)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 7 (11)
White blood cell decreased (Investigations) | 28 (107)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-14): https://cdn.clinicaltrials.gov/large-docs/02/NCT03159702/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/02/NCT03159702/ICF_001.pdf